CLINICAL TRIAL: NCT04923373
Title: Early Function Recovery in Geriatric Patients With Total Knee Arthroplasty by Telerehabilitation
Brief Title: Telerehabilitation After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Drzał-Grabiec, Professor, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/11/2006
Record Dates: First submitted 2021-05-25; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Telerehabilitation; Total Knee Arthoplasty; Physiotherapy
Keywords: disability; geriatric
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The patients (n=105) were randomly divided into two groups: telerehabilitation group (n=54) - 42 women and 12 men and control group (n=51) 40 women and 11 men - direct physiotherapist supervised group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telerehabilitation (Experimental): physiotherapeutic programme brochure exercises 7/week controlled by phone every week (5x in total)
  Interventions: Other: telerehabilitation
- standard physiotherapy (Active Comparator): Supervised physical therapy 3/ week,
  + physiotherapeutic programme brochure 4/week
  Interventions: Procedure: standard physiotherapy

INTERVENTIONS:
Other: telerehabilitation — Procedure for both groups:
  I pre surgery evaluation
  1. initial training in hospital
  2. physiotherapeutic programme telerehabilitation versus standard 7 times a week
  Therapy duration: 6 weeks post-surgery II 6weeks post-surgery evaluation
  Arms: telerehabilitation
Procedure: standard physiotherapy — standard physiotherapy
  Arms: standard physiotherapy

SUMMARY:
The aim of this study was to assess the function, pain intensity and walking distance in patients prior to and after total knee arthroplasty, who received therapy either in a clinic under direct supervision of a physical therapist and patients who received telerehabilitation.

DETAILED DESCRIPTION:
The study population consisted of 105 patients who had knee arthroplasty due to knee arthrosis followed by 6- weeks physiotherapy, mean age 68.5 ± 7.3 years. The patients were randomly divided into two groups: I - telerehabilitation group (n=54), and II clinical control group (n=51), who received physiotherapy supervised by physiotherapist. All patients were given the following tests: VAS (0-10), 6-Minute Walk Test, and KSS - Knee Society Score.

ELIGIBILITY:
Inclusion Criteria:

* total cemented knee arthroplasty with posterior stability (PS -cruciate sacrificing, posterior stabilized),
* informed consent to participate in the study,
* full medical record,
* patients' regular control visits,
* knee degenerative disorder stage II and III according to Altman classification,
* ability to understand and independently perform the complete physiotherapeutic programme

Exclusion Criteria:

* partial arthroplasty,
* deformation aetiology other knee degenerative disorder,
* cognitive disorders resulting in inability to fill out the study questionnaire, - degenerative disorders of multiple joints,
* poor general health that prevented the patient from understanding or performing the full physiotherapeutic programme,
* intraoperative and postoperative complications preventing the patient from understanding or performing the full physiotherapeutic programme,
* lack of informed consent to participate in the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

PRIMARY OUTCOMES:
Change in 6 - Minute Walk Test | Change from baseline- 1st measurement before total knee arthroplasty and final - 2nd measurement in 6 weeks after total knee arthroplasty and physiotherapy
  Change in walking distance in 6 minutes ( in meters)
Change in Knee Society Score | Change from baseline- 1st measurement before total knee arthroplasty and final - 2nd measurement in 6 weeks after total knee arthroplasty and physiotherapy
  Change in disability measured by Knee disability score (min 0 - max 200 points). Higher scores mean a better outcome.
Change in range of knee motion [degrees] | Change from baseline- 1st measurement before total knee arthroplasty and final - 2nd measurement in 6 weeks after total knee arthroplasty and physiotherapy
  Change in knee flexion
Change of knee pain intensity in Visual Analogue Scale | Change from baseline- 1st measurement before total knee arthroplasty and final - 2nd measurement in 6 weeks after total knee arthroplasty and physiotherapy
  Change of knee pain intensity (0-10), 0 - no pain, 10 - worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Szpital Specjalistyczny im. Świętej Rodziny, Rudna Mała, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Truszczynska-Baszak A, Dadura E, Drzal-Grabiec J, Tarnowski A. Static balance assessment in patients with severe osteoarthritis of the knee. Knee. 2020 Oct;27(5):1349-1356. doi: 10.1016/j.knee.2020.06.014. Epub 2020 Jul 27. PMID 33010747
- [Result] Benz T, Angst F, Oesch P, Hilfiker R, Lehmann S, Mueller Mebes C, Kramer E, Verra ML. Comparison of patients in three different rehabilitation settings after knee or hip arthroplasty: a natural observational, prospective study. BMC Musculoskelet Disord. 2015 Oct 24;16:317. doi: 10.1186/s12891-015-0780-2. PMID 26497597
- [Result] Russell TG, Buttrum P, Wootton R, Jull GA. Rehabilitation after total knee replacement via low-bandwidth telemedicine: the patient and therapist experience. J Telemed Telecare. 2004;10 Suppl 1:85-7. doi: 10.1258/1357633042614384. PMID 15603622
- [Result] Piqueras M, Marco E, Coll M, Escalada F, Ballester A, Cinca C, Belmonte R, Muniesa JM. Effectiveness of an interactive virtual telerehabilitation system in patients after total knee arthoplasty: a randomized controlled trial. J Rehabil Med. 2013 Apr;45(4):392-6. doi: 10.2340/16501977-1119. PMID 23474735
- [Result] Moffet H, Tousignant M, Nadeau S, Merette C, Boissy P, Corriveau H, Marquis F, Cabana F, Ranger P, Belzile EL, Dimentberg R. In-Home Telerehabilitation Compared with Face-to-Face Rehabilitation After Total Knee Arthroplasty: A Noninferiority Randomized Controlled Trial. J Bone Joint Surg Am. 2015 Jul 15;97(14):1129-41. doi: 10.2106/JBJS.N.01066. PMID 26178888